CLINICAL TRIAL: NCT05412641
Title: Evaluation of the FELLAS Responsible Fatherhood Project
Acronym: FELLAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Partnership for Maternal & Child Health of Northern New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FELLAS project
Record Dates: First submitted 2022-04-25; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-04

CONDITIONS: Responsible Fatherhood

STUDY DESIGN:
Intervention Model Description: Fathers participate in and educational program designed to help them improve (1) healthy marriage/relationship skills, (2) conflict resolution skills, (3) financial management/economic stability, and (4) parenting skills.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention - Responsible Fatherhood Programming (Other): Participants receive educational programming to include: 24/7 Dad, Couples Communication I, and a comprehensive program targeting financial literacy/money management. The study features only one group. Participants will receive the intervention described. There is no control group.
  Interventions: Other: Intervention - Responsible Fatherhood Programming

INTERVENTIONS:
Other: Intervention - Responsible Fatherhood Programming — Participants receive educational programming to include: 24/7 Dad, Couples Communication I, and a comprehensive program targeting financial literacy/money management.

SUMMARY:
The Partnership for Maternal and Child Health of Northern New Jersey, Inc. (PMCH) is implementing a fatherhood project with the goal of strengthening father-child engagement, improving economic stability, and improving healthy marriage/relationship skills among participants. FELLAS serves community-based fathers 18 years of age or older who reside in Essex County, New Jersey and have at least one child under the age of 24. The program model has three components: to improve responsible parenting using 24/7 Dad, an evidence based curriculum; to improve healthy marriage/relationship skills using Couple Communication I, an evidence based relationship and marriage strengthening curriculum that includes home visits; and to improve economic stability using a comprehensive array of services designed to provide an employment assessment, strengthen basic technology skills, and strengthen pre-employment soft skills. Evaluation activities include a self-report questionnaire administered (1) immediately prior to beginning the program (pretest), (2) immediately after completion of the program (posttest), and (3) six months after the posttest. Focus groups will also provide qualitative data concerning the effects of the program.

DETAILED DESCRIPTION:
The Partnership for Maternal and Child Health of Northern New Jersey, Inc. (PMCH) is implementing a fatherhood project with the goal of strengthening father-child engagement, improving economic stability, and improving healthy marriage/relationship skills among participants. FELLAS serves community-based fathers 18 years of age or older who reside in Essex County, New Jersey and have at least one child under the age of 24.

The program model has three components: to improve responsible parenting using 24/7 Dad, an evidence based curriculum; to improve healthy marriage/relationship skills using Couple Communication I, an evidence based relationship and marriage strengthening curriculum that includes home visits; and to improve economic stability using a comprehensive array of services designed to provide an employment assessment, strengthen basic technology skills, and strengthen pre-employment soft skills.

The Theory of Change the investigators will use in this project is the Health Belief Model (HBM). According to the HBM, individuals are most likely to make behavior changes when they believe that a problem is potentially severe, they are personally susceptible to the problem, the benefits to making change outweigh the challenges or risk, and they believe that they can, in fact, make the desired changes.

The four primary research questions deal with: 1) communication and empathy skills toward one's partner; 2) conflict resolution skills and associated behavior patterns; 3) financial management and economic stability; 4) positive effective parenting skills. The investigators have selected these research questions because the investigators believe, and the literature supports the position, that these factors are of major importance in becoming an actively engaged and responsible father.

The research evidence is clear. Children who do not have a responsible father in their lives suffer several negative outcomes when compared to children who do have a responsible father in their lives. Following the HBM, the approach the investigators will take in delivering the intervention will be to emphasize the importance of fatherhood engagement in the lives of their children and:

1. how the lack of father engagement can result in serious negative outcomes for their children relative to child development - and on into adulthood (severity);
2. if they are not personally, actively engaged in the lives of their children, then their children are also likely to experience serious negative outcomes (susceptibility);
3. though being an actively involved, responsible father is not easy, the results, both for their children and themselves will be worth the effort (benefits vs challenge);
4. becoming an actively involved, responsible father is a difficult task, but it is something the participants can do; and the FELLAS project is here to help (self-efficacy).

Evaluation activities include a self-report questionnaire administered (1) immediately prior to beginning the program (pretest), (2) immediately after completion of the program (posttest), and (3) six months after the posttest. Focus groups will also provide qualitative data concerning the effects of the program.

The investigators hypothesize that following the intervention, the participants will show improvement in:

(1) communication and empathy skills toward their partner; (2) conflict resolution skills and associated behavior patterns; (3) financial management and economic stability; (4) positive effective parenting scores.

ELIGIBILITY:
Inclusion Criteria: Must be a father, have at least one child 24 years old or younger, and reside in Essex County, New Jersey.

-

Exclusion Criteria: Not a father, or a father with all children older than 24, not a resident of Essex County, New Jersey

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the inclusion criteria include the requirement that participants be fathers, one could assume that all participants will be male. If, however, a transgender female is a father, then she would be eligible to participate in the study.
Enrollment: 540 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Communication skills | From pretest to posttest; approximately five weeks
  Participants will improve scores on healthy marriage/relationship skills.The outcome, Healthy marriage/relationship skills is measured using a 13 item scale. A sample item is: "Before criticizing my partner' I try to imagine how I would feel if I were in her place." Each item is scored on a five point response option from 1 (does not describe me well) to 5 (describes me very well).
Communication skills at follow-up | Pretest to six-month followup
  Participants will improve scores on healthy marriage/relationship skills.The outcome, Healthy marriage/relationship skills is measured using a 13 item scale. A sample item is: "Before criticizing my partner' I try to imagine how I would feel if I were in her place." Each item is scored on a five point response option from 1 (does not describe me well) to 5 (describes me very well).
Conflict resolution skills | From pretest to posttest; approximately five weeks
  Participants will improve scores on conflict resolution skills. The outcome conflict resolution sills is measured by using a six item scale. A sample items is: "I take time to relax before I bring up a problem." Each item is scored on a four point response option from 1 (strongly disagree) to 4 (strongly agree).
Conflict resolution skills at follow-up | Pretest to six-month followup
  Participants will improve scores on conflict resolution skills. The outcome conflict resolution sills is measured by using a six item scale. A sample items is: "I take time to relax before I bring up a problem." Each item is scored on a four point response option from 1 (strongly disagree) to 4 (strongly agree).
Economic stability skills | From pretest to posttest; approximately five weeks
  Participants will improve scores on economic stability skills. The outcome, Economic stability skills is measure by using a six item scale. A sample item is: "Learning how to budget is a useful way to manage money and reach goals." Each item is scored on a four point response option from 1 (strongly disagree) to 4 (strongly agree).
Economic stability skills at follow-up | From pretest to six month follow-up/
  Participants will improve scores on economic stability skills. The outcome, Economic stability skills is measure by using a six item scale. A sample item is: "Learning how to budget is a useful way to manage money and reach goals." Each item is scored on a four point response option from 1 (strongly disagree) to 4 (strongly agree).
Improved Parenting Skills | From pretest to posttest; approximately five weeks
  Participants will improve in parenting skills. The outcome, Improved Parenting Skills, is measured using a 12 item scale. A sample item is: "Set and stick to reasonable limits and rules. Each item is scored on a seven point response option from 0 (low skills) to 6 (high skills).
Improved Parenting Skills at follow-up | From pretest to six month follow-up.
  Participants will improve in parenting skills. The outcome, Improved Parenting Skills, is measured using a 12 item scale. A sample item is: "Set and stick to reasonable limits and rules. Each item is scored on a seven point response option from 0 (low skills) to 6 (high skills).

CONTACTS AND LOCATIONS:
Locations (1):
- Partnership for Maternal & Child Health of Northern New Jersey, Newark, New Jersey, United States